CLINICAL TRIAL: NCT06880874
Title: A Clinical Study to Evaluate the Relative Bioavailability of Enlicitide Formulations in Healthy Adult Participants
Brief Title: A Clinical Study to Evaluate Enlicitide (MK-0616) Formulations in Healthy Adult Participants (MK-0616-035)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-035; MK-0616-035 (Other: MSD)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: enlicitide reference tablet (Experimental): Participants receive a single oral dose of enlicitide reference tablet.
  Interventions: Drug: Enlicitide
- Treatment B: enlicitide test tablet (Experimental): Participants receive a single oral dose of enlicitide test tablet.
  Interventions: Drug: Enlicitide

INTERVENTIONS:
Drug: Enlicitide — Oral Tablet
  Other Names: MK-0616; enlicitide decanoate

SUMMARY:
The goal of the study is to learn what happens to different forms of enlicitide medications in a healthy person's body over time. Researchers will compare the amount of enlicitide in the healthy person's body over time when enlicitide is given in different formulations.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior
* Has body mass index (BMI) ≥18 kg/m^2 and ≤32 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of gastrointestinal disease which may affect food and drug absorption or has had a gastric bypass or similar surgery
* Has history of cancer (malignancy)
* Has positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the AUC0-24hr of enlicitide.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-Last of enlicitide.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-Inf of enlicitide.
Maximum Plasma Concentration (Cmax) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Blood samples will be collected to determine the Cmax of enlicitide.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 8 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com